CLINICAL TRIAL: NCT04026048
Title: A Randomized Controlled Trial of Online Cognitive Behavior Therapy for Insomnia (CBT-I) and Perceived Cognitive Impairment (PCI) in Cancer Survivors
Brief Title: Online Treatment of Cognitive Impairment and Insomnia in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Sheila Garland, Associate Professor of Psychology and Oncology at Memorial University of Newfoundland, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200427; PJT 162428 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2019-07-04; First posted 2019-07-19 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Insomnia; Cognitive Impairment
Keywords: Cognitive Behaviour Therapy for Insomnia; CBT-I; Cancer; Insomnia; Sleep; Perceived Cognitive Impairment
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders; Cognitive Dysfunction | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behaviour Therapy for Insomnia (CBT-I) (Experimental): Participants will receive individualized CBT-I delivered by video-conferencing over the course of eight weeks.
  Interventions: Behavioral: Cognitive Behaviour Therapy for Insomnia (CBT-I)
- Waitlist Control Group (Experimental): Participants in the waitlist control group will be required to monitor their sleep with sleep diaries for 7 weeks. They will receive CBT-I delivered by video-conferencing immediately after the waiting period.
  Interventions: Behavioral: Cognitive Behaviour Therapy for Insomnia (CBT-I)

INTERVENTIONS:
Behavioral: Cognitive Behaviour Therapy for Insomnia (CBT-I) — CBT-I is a manualized multi-component intervention that includes sleep restriction, stimulus control, cognitive restructuring, relaxation training, and sleep hygiene.

SUMMARY:
The investigators will answer the question of whether treating insomnia using Cognitive Behavior Therapy for Insomnia (CBT-I) can improve perceived cognitive impairment (PCI) in cancer survivors compared to a waitlist control group. The investigators will recruit 124 people with insomnia and cognitive complaints who have completed cancer treatment at least 6 months prior to the study.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial of immediate treatment with CBT-I compared to a delayed treatment group with 124 cancer survivors who have completed primary treatment at least 6 months prior and report PCI and insomnia. Participants who are randomized to the immediate treatment group will receive CBT-I over the course of seven weekly one hour sessions, after which the delayed treatment group will receive the intervention. Both groups will complete follow up assessments three and six months after completing treatment. PCI will be assessed using the Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) as the primary outcome. To provide an objective assessment of cognition, the investigators have included the neurocognitive measures recommended by the International Cognition and Cancer Task Force. Other measures will include fatigue, anxiety, depression, and work productivity.

The investigators hypothesize that the online CBT-I group will report significantly greater improvements in perceived cognitive function compared to the waitlist control immediately post-treatment (primary endpoint). The investigators also hypothesize that these improvements will be maintained up at 6-months follow up (secondary endpoint).

ELIGIBILITY:
Inclusion Criteria for individuals with non-hematological malignancies:

* Men and women who are easily able to understand and read English
* No current evidence of cancer or clinically stable/inactive disease
* Received and completed all adjuvant treatments at least 6 months prior to study entry to allow for neural stabilization and recovery
* Self-reported PCI as indicated by a score of "sometimes" or higher ("quite a lot" or "always") on at least two out of three questions that assess memory, concentration, and attention
* Meet the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for insomnia disorder and have a score of 8 or greater on the Insomnia Severity Index (ISI)
* Have good performance status as indicated by an Eastern Cooperative Oncology Group (ECOG) score of 0-2
* Have high-speed internet connection, webcam, and are fluent using the internet

Inclusion Criteria for individuals with hematological malignancies:

* Men and women who are easily able to understand and read English
* A diagnosis of a hematological malignancy currently in remission
* Completed cancer treatments including transplant, chemotherapy and/or immunotherapy at least 6 months prior to study entry
* Self-reported PCI as indicated by a score of "sometimes" or higher ("quite a lot" or "always") on at least two out of three questions that assess memory, concentration, and attention
* Meet the DSM-5 criteria for insomnia disorder and have a score of 8 or greater on the Insomnia Severity Index
* Have good performance status as indicated by an ECOG score of 0-2
* Have high-speed internet connection, webcam, and are fluent using the internet

Exclusion Criteria for individuals with and without hematological malignancies:

* Another sleep disorder, besides insomnia, that is not adequately treated (ie: untreated obstructive sleep apnea)
* The presence of another psychological disorder that is not currently stable and/or would impair the ability to participate in the study
* A major sensory deficit (e.g. blindness)
* A neurologic or major medical condition known to affect cognitive function (e.g., Parkinson's)
* A history of cranial radiation
* A history of any other condition that may affect cognitive functioning (e.g., traumatic brain injury)
* Previous experience with CBT-I

Other considerations:

* Participants will not be excluded for using psychotropic medication prior to study entry (e.g. antidepressants) provided that the dose was not recently altered (stable over the previous 6 weeks)
* Considering the potential for prescription of medications to help with sleep (e.g. hypnotics, sedatives, and antidepressants) within the cancer population, medication use throughout the study will be tracked and adjusted for in the statistical analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila N Garland, PhD, Principal Investigator — Memorial University of Newfoundland
Locations (1):
- Memorial University of Newfoundland, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811
- [Derived] Greeley KM, Lee RM, Tulk J, Harding SV, Yi Y, Aubrey-Bassler K, Garland SN. Recording and reporting of adverse events during a randomized controlled trial of cognitive behavioural therapy for insomnia (CBT-I) among cancer survivors. Sleep Sci Pract. 2025;9(1):10. doi: 10.1186/s41606-025-00129-8. Epub 2025 May 10. PMID 40352744
- [Derived] Greeley KM, Rash J, Tulk J, Savard J, Seal M, Urquhart R, Thoms J, Laing K, Fawcett E, Garland SN. Factors associated with significant improvement in cancer-related fatigue after completing cognitive behavioral therapy for insomnia in cancer survivors. Support Care Cancer. 2025 Apr 28;33(5):432. doi: 10.1007/s00520-025-09482-x. PMID 40295384
- [Derived] Greeley KM, Rash J, Tulk J, Savard J, Seal M, Urquhart R, Thoms J, Laing K, Fawcett E, Garland SN. Impact and mechanisms of cognitive behavioral therapy for insomnia on fatigue among cancer survivors: a secondary analysis of a randomized controlled trial. Sleep. 2025 Jun 13;48(6):zsaf014. doi: 10.1093/sleep/zsaf014. PMID 39826090
- [Derived] Garland SN, Tulk J, Savard J, Rash JA, Browne S, Urquhart R, Seal M, Thoms J, Laing K. Randomized Controlled Trial of Virtually Delivered Cognitive Behavioral Therapy for Insomnia to Address Perceived Cancer-Related Cognitive Impairment in Cancer Survivors. J Clin Oncol. 2024 Jun 10;42(17):2094-2104. doi: 10.1200/JCO.23.02330. Epub 2024 Mar 29. PMID 38552188

RESULTS

PARTICIPANT FLOW:
Period: Pre-treatment to Treatment Completion
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
Started | 63 | 69
Completed | 58 | 63
Not Completed | 5 | 6
Period: 3 Month Follow-up
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
Started | 58 | 63
Completed | 55 | 60
Not Completed | 3 | 3
Period: 6 Month Follow-up
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
Started | 55 | 60
Completed | 53 | 59
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group | Total
Number analyzed (Participants) | 63 | 69 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.21 (11.93) | 61.25 (10.60) | 60.28 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 52 | 102
  Male | 13 | 17 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 57 | 65 | 122
  BIPOC | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  Canada | 63 | 69 | 132
Years of education [Count of Participants; unit: Participants]
  High school (≤11 years) | 4 | 2 | 6
  College (12-14 years) | 18 | 24 | 42
  Postsecondary (≥15 years) | 41 | 43 | 84
Employment status [Count of Participants; unit: Participants]
  Not working/retired | 36 | 48 | 84
  Working (part or full-time) | 27 | 21 | 48
Cancer type [Count of Participants; unit: Participants]
  Breast | 25 | 29 | 54
  Prostate and male genitourinary | 2 | 5 | 7
  Female genitourinary | 6 | 5 | 11
  GI tract | 2 | 5 | 7
  Hematologic | 11 | 5 | 16
  Skin | 2 | 6 | 8
  Other | 4 | 2 | 6
  Multiple types | 11 | 12 | 23
Time since cancer diagnosis (years) [Count of Participants; unit: Participants]
  <2 | 7 | 7 | 14
  2-4 | 11 | 21 | 32
  5-9 | 17 | 14 | 31
  ≥10 | 28 | 26 | 54
Cancer stage [Count of Participants; unit: Participants] — Cancer stage was determined at time of diagnosis. Generally, a greater stage indicates worse outcomes.
  Stage 0 - carcinoma in situ, a precancerous change; Stage 1 - the tumour is usually small and hasn't grown outside of the organ it started in; Stages 2 and 3 - the tumour is larger or has grown outside of the organ it started in to nearby tissue; Stage 4 - the cancer has spread through the blood or lymphatic system to another part of the body.
  Participants
    Stage 0/in situ | 1 | 3 | 4
    Stage I | 12 | 15 | 27
    Stage II | 13 | 10 | 23
    Stage III | 15 | 13 | 28
    Stage IV | 2 | 5 | 7
    Unknown/not applicable | 20 | 23 | 43
Cancer treatments received [Count of Participants; unit: Participants]
  Surgery | 52 | 65 | 117
  Chemotherapy | 46 | 35 | 81
  Radiation | 38 | 38 | 76
  Hormone therapy | 13 | 29 | 42
  Other | 4 | 4 | 8
Time since insomnia began (months) [Mean (Standard Deviation); unit: months] | 99.19 (71.17) | 88.56 (79.23) | 93.63 (75.39)
Baseline insomnia score [Mean (Standard Deviation); unit: units on a scale] — The Insomnia Severity Index (ISI) is a 7-item measure that assesses the severity of insomnia symptoms over the past 7 days. Responses can range from 0 to 4, where higher scores indicate more acute symptoms of insomnia.
  A total score of 0-7 indicates "no clinically significant insomnia," 8-14 means "subthreshold insomnia," 15-21 is "clinical insomnia (moderate severity)," and 22-28 means "clinical insomnia (severe)."
  units on a scale | 17.27 (3.53) | 17.88 (3.83) | 17.59 (3.69)
Baseline perceived cognitive impairment score [Mean (Standard Deviation); unit: units on a scale] — The Functional Assessment of Cancer Therapy -Cognitive Function (FACT-Cog) scale contains 37 items to measure Perceived Cognitive Impairments (PCI), Impact of Perceived Cognitive Impairments on QoL, Comments from Others, Perceived Cognitive Abilities.
  Responses range from 0, ''never,'' to 4, ''several times a day,'' in the previous 7 days and negatively worded items are reverse scored to create subscale scores. Scores on the PCI subscale can range from 0 to 72 points (negatively worded items are reverse coded), with a higher score indicative of better self-reported cognitive functioning.
  units on a scale | 39.40 (12.32) | 38.80 (13.86) | 39.1 (13.10)

OUTCOME MEASURES:

1. Primary Outcome: The Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) Version 3
Description: The FACT-Cog was used to measure perceived cognitive impairment (PCI). It is a 37-item questionnaire with four cognitive subscales: perceived cognitive impairments, impact on quality of life, comments from others, and perceived cognitive abilities. Responses range from 0, ''never,'' to 4, ''several times a day,'' in the previous 7 days and negatively worded items are reverse scored to create subscale scores. Scores on the PCI subscale can range from 0 to 72 points, with a higher score indicative of better self-reported cognitive functioning and quality of life. A change of 5.9-points has been established as clinically meaningful change on the FACT-Cog PCI subscale
Time Frame: Change from Baseline to Week 4, Week 8, 3 month follow up, 6 month follow up
Population: Although there were 63 and 69 participants who began treatment in the CBT-I and waitlist groups, respectively, we only have data from participants whose data were complete for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
Number analyzed (Participants) | 63 | 69
score on a scale
  Baseline | 39.39 (12.32) | 38.79 (13.85)
  4 weeks: number analyzed (Participants) | 60 | 68
  4 weeks | 48.28 (11.89) | 44.71 (13.84)
  8 weeks: number analyzed (Participants) | 59 | 67
  8 weeks | 53.44 (12.01) | 43.00 (12.89)
  3 months follow-up: number analyzed (Participants) | 55 | 66
  3 months follow-up | 53.16 (11.37) | 46.21 (19.64)
  6 months follow-up: number analyzed (Participants) | 53 | 59
  6 months follow-up | 52.47 (12.89) | 51.46 (14.10)

2. Secondary Outcome: The Insomnia Severity Index (ISI)
Description: The ISI is designed to specifically assess the severity of insomnia symptoms, the impact on daytime functioning, and the amount of associated distress. The ISI has 7 questions, which are summed to compute a total score. The range of the ISI is 0-28 with the higher the value, the more severe the insomnia severity.
Time Frame: Change from Baseline to Week 4, Week 8, 3 month follow up, 6 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on Insomnai Severity Index
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
Number analyzed (Participants) | 63 | 69
score on Insomnai Severity Index
  Basline: number analyzed (Participants) | 63 | 67
  Basline | 17.27 (3.53) | 15.06 (4.57)
  4 weeks: number analyzed (Participants) | 60 | 63
  4 weeks | 9.67 (4.01) | 9.77 (4.81)
  8 weeks: number analyzed (Participants) | 57 | 64
  8 weeks | 6.03 (3.90) | 6.34 (4.30)
  3 months follow-up: number analyzed (Participants) | 54 | 58
  3 months follow-up | 7.11 (4.84) | 6.37 (4.60)
  6 months follow-up: number analyzed (Participants) | 51 | 57
  6 months follow-up | 7.94 (5.60) | 6.28 (4.23)

3. Secondary Outcome: Sleep Efficiency Measured by The Consensus Sleep Diary (CSD)
Description: Sleep efficiency is the percentage of time spent asleep while in bed. It is calculated by dividing the amount of time spent asleep (in minutes) by the total amount of time in bed (in minutes). The unit of measure is a percentage and is averaged over the whole week for the total sleep efficiency score.
Time Frame: Change from Baseline to Week 4, Week 8, 3 month follow up, 6 month follow up
Population: Although there were 63 and 69 participants who began treatment in the CBT-I and waitlist groups, respectively, we only have data from participants whose consensus sleep diaries were complete and returned.
Measure: Mean (Standard Deviation); unit: percentage of sleep efficiency
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
Number analyzed (Participants) | 63 | 69
percentage of sleep efficiency
  Baseline: number analyzed (Participants) | 63 | 66
  Baseline | 73.22 (12.45) | 74.03 (13.58)
  4 weeks: number analyzed (Participants) | 60 | 63
  4 weeks | 87.18 (8.17) | 88.10 (6.24)
  8 weeks: number analyzed (Participants) | 56 | 63
  8 weeks | 89.63 (7.10) | 89.33 (6.41)
  3 month follow-up: number analyzed (Participants) | 50 | 54
  3 month follow-up | 88.58 (8.02) | 87.22 (7.62)
  6 month follow-up: number analyzed (Participants) | 48 | 54
  6 month follow-up | 88.52 (7.88) | 87.83 (6.81)

4. Secondary Outcome: Sleep-onset Latency Measured by The Consensus Sleep Diary (CSD)
Description: The sleep diary will be used to calculate sleep-onset latency, which is the length of time that it takes to accomplish the transition from full wakefulness to sleep. The unit of measure is minutes and is averaged over the whole week for the total sleep onset latency score.
Time Frame: Change from Baseline to Week 4, Week 8, 3 month follow up, 6 month follow up
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
Number analyzed (Participants) | 63 | 69
minutes
  Baseline: number analyzed (Participants) | 63 | 66
  Baseline | 40.56 (32.40) | 41.48 (34.22)
  4 weeks: number analyzed (Participants) | 60 | 63
  4 weeks | 16.68 (15.73) | 16.98 (13.43)
  8 weeks: number analyzed (Participants) | 56 | 63
  8 weeks | 12.68 (8.98) | 15.41 (11.7)
  3 month follow-up: number analyzed (Participants) | 50 | 54
  3 month follow-up | 16.70 (18.44) | 21.43 (16.04)
  6 month follow-up: number analyzed (Participants) | 48 | 54
  6 month follow-up | 14.71 (10.41) | 22.26 (20.24)

5. Secondary Outcome: Wake After Sleep Onset Measured by The Consensus Sleep Diary (CSD)
Description: The sleep diary will be used to calculate wake after sleep onset, which refers to periods of wakefulness occurring after defined sleep onset. The score is reported in minutes and is averaged over the whole week for the total wake after sleep onset.
Time Frame: Change from Baseline to Week 4, Week 8, 3 month follow up, 6 month follow up
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
Number analyzed (Participants) | 63 | 69
minutes
  Baseline: number analyzed (Participants) | 63 | 66
  Baseline | 63.29 (41.99) | 50.80 (34.14)
  4 weeks: number analyzed (Participants) | 60 | 63
  4 weeks | 23.32 (17.30) | 19.90 (14.87)
  8 weeks: number analyzed (Participants) | 56 | 63
  8 weeks | 21.84 (19.80) | 20.06 (18.95)
  3 month follow-up: number analyzed (Participants) | 50 | 54
  3 month follow-up | 20.06 (20.46) | 22.87 (19.86)
  6 month follow-up: number analyzed (Participants) | 48 | 54
  6 month follow-up | 21.46 (20.24) | 21.85 (20.34)

6. Secondary Outcome: Total Sleep Time Measured by The Consensus Sleep Diary (CSD):
Description: The sleep diary will be used to calculate total sleep time. The score is reported in minutes and is averaged over the whole week for the total sleep time.
Time Frame: Change from Baseline to Week 4, Week 8, 3 month follow up, 6 month follow up
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
Number analyzed (Participants) | 63 | 69
minutes
  Baseline: number analyzed (Participants) | 63 | 66
  Baseline | 370.06 (67.72) | 378.41 (81.09)
  4 weeks: number analyzed (Participants) | 60 | 63
  4 weeks | 358.77 (64.05) | 376.08 (59.71)
  8 weeks: number analyzed (Participants) | 56 | 63
  8 weeks | 392.14 (52.52) | 406.40 (57.11)
  3 month follow-up: number analyzed (Participants) | 50 | 54
  3 month follow-up | 412.06 (68.69) | 418.81 (62.12)
  6 month follow-up: number analyzed (Participants) | 48 | 54
  6 month follow-up | 401.42 (84.67) | 429.24 (56.60)

7. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: Anxiety and Depression will be measured using the HADS, which is a 14-item, self-rated instrument for anxiety (7 items) and depression (7 items) symptoms in the past week and has been extensively used in people with cancer. Scores range from 0-21 with below 7 indicating a non-case and the higher the score indicates greater symptom severity.
Time Frame: Change from Baseline to Week 4, Week 8, 3 month follow up, 6 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
Number analyzed (Participants) | 63 | 69
score on a scale
  Baseline depression: number analyzed (Participants) | 63 | 67
  Baseline depression | 7.90 (2.88) | 6.39 (3.72)
  4 weeks depression: number analyzed (Participants) | 60 | 63
  4 weeks depression | 4.45 (3.48) | 4.63 (3.65)
  8 weeks depression: number analyzed (Participants) | 57 | 64
  8 weeks depression | 3.14 (3.29) | 3.09 (3.14)
  3 month follow-up depression: number analyzed (Participants) | 54 | 58
  3 month follow-up depression | 3.57 (2.88) | 5.90 (2.36)
  6 month follow-up depression: number analyzed (Participants) | 51 | 57
  6 month follow-up depression | 4.24 (3.52) | 3.30 (2.99)
  Baseline anxiety: number analyzed (Participants) | 63 | 67
  Baseline anxiety | 9.33 (3.48) | 8.70 (4.24)
  4 weeks anxiety: number analyzed (Participants) | 60 | 63
  4 weeks anxiety | 6.88 (3.25) | 7.97 (3.78)
  8 weeks anxiety: number analyzed (Participants) | 57 | 64
  8 weeks anxiety | 5.89 (3.31) | 7.08 (4.47)
  3 month follow-up anxiety: number analyzed (Participants) | 54 | 58
  3 month follow-up anxiety | 6.04 (3.79) | 5.97 (4.41)
  6 month follow-up anxiety: number analyzed (Participants) | 51 | 57
  6 month follow-up anxiety | 6.18 (4.33) | 5.67 (3.82)

8. Secondary Outcome: Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF)
Description: Fatigue will be measured using the Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF), which is a 30 item self-report measure comprised of five subscales (general, emotional, physical, mental, vigor) and a total fatigue score. Each subscale score ranges from 0 to 24. The Total MSFI-SF score is calculated by adding the general, physical, emotional and mental subscale scores and subtracting vigor subscale score. Total MFSI-SF score ranges from -24 to 96 with a higher score indicating higher levels of cancer-related fatigue experienced by the patient.
Time Frame: Change from Baseline to Week 4, Week 8, 3 month follow up, 6 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
Number analyzed (Participants) | 63 | 69
score on a scale
  Baseline: number analyzed (Participants) | 63 | 67
  Baseline | 29.57 (16.75) | 26.64 (19.38)
  4 weeks: number analyzed (Participants) | 63 | 63
  4 weeks | 16.52 (17.50) | 17.17 (20.49)
  8 weeks: number analyzed (Participants) | 63 | 64
  8 weeks | 4.72 (16.17) | 6.05 (19.62)
  3 month follow-up: number analyzed (Participants) | 63 | 58
  3 month follow-up | 9.13 (16.44) | 6.79 (18.41)
  6 month follow-up: number analyzed (Participants) | 63 | 57
  6 month follow-up | 10.04 (18.13) | 5.95 (17.65)

9. Secondary Outcome: The Hopkins Verbal Learning Test-Revised (HVLT-R)
Description: The Hopkins Verbal Learning Test-Revised (HVLT-R) is a brief assessment of verbal learning and memory (immediate recall, delayed recall, delayed recognition). When scoring the HVLT-R, the three learning trials are combined to calculate a total recall score; the delayed recall trial creates the delayed recall score; the retention (%) score is calculated by dividing the delayed recall trial by the higher of learning trial 2 or 3; and the recognition discrimination index is comprised by subtracting the total number of false positives from the total number of true positives. These scores are then converted to an age-based T score (Mean=50, SD=10). Higher scores represent better verbal learning and memory.
Time Frame: Change from Baseline to Week 8, 3 month follow up, 6 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t score
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
Number analyzed (Participants) | 63 | 69
t score
  Baseline: number analyzed (Participants) | 63 | 67
  Baseline | 49.84 (10.72) | 49.22 (12.64)
  8 weeks: number analyzed (Participants) | 55 | 64
  8 weeks | 49.11 (11.63) | 50.19 (10.95)
  3 month follow-up: number analyzed (Participants) | 51 | 59
  3 month follow-up | 54.25 (9.66) | 53.36 (11.47)
  6 month follow-up: number analyzed (Participants) | 48 | 54
  6 month follow-up | 55.94 (10.67) | 54.54 (10.94)

10. Secondary Outcome: The Controlled Oral Word Association Test (COWAT)
Description: The COWAT is a measure of verbal fluency, cognitive and motor speed, cognitive flexibility, strategy utilization, suppression of interference, and response inhibition. The total score is the total number of different words produced for all three letters in a timeframe of 3 minutes (1 minute for each letter). The scores are adjusted based on age and education level. A greater score indicates better verbal fluency. A score less then 33 indicates below average performance, scores between 34 and 45 indicate average performance, and scores greater than 45 are above average, with scores greater than 52 indicate superior performance. A minimum score is 0 (no words produced) and there is no set maximum score, as it depends on how many words can be produced in the given time frame.
Time Frame: Change from Baseline to Week 8, 3 month follow up, 6 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: adj score on a scale
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
Number analyzed (Participants) | 63 | 69
adj score on a scale
  Baseline: number analyzed (Participants) | 63 | 66
  Baseline | 47.14 (11.48) | 44.41 (12.31)
  8 weeks: number analyzed (Participants) | 57 | 62
  8 weeks | 46.77 (11.12) | 47.50 (13.61)
  3 month follow-up: number analyzed (Participants) | 52 | 59
  3 month follow-up | 51.04 (12.91) | 48.42 (12.20)
  6 month follow-up: number analyzed (Participants) | 47 | 53
  6 month follow-up | 50.02 (11.44) | 49.62 (13.87)

11. Secondary Outcome: The Digit Span
Description: The Digit Span test is a subtest of both the Wechsler Adult Intelligence Scale (WAIS) and the Wechsler Memory Scale (WMS). Part A of digit span (the forward span) captures attention efficiency and capacity, and part B (the backward span) is an executive task dependent on working memory. The Digit Span subtest will be scored as one summary value. The unit of measure is the total recall. Scores on this measure range from 0-48, where greater scores indicates greater attention efficiency, capacity and working memory.
Time Frame: Change from Baseline to Week 8, 3 month follow up, 6 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
Number analyzed (Participants) | 63 | 69
score on a scale
  Baseline: number analyzed (Participants) | 63 | 66
  Baseline | 28.49 (4.06) | 28.44 (5.03)
  8 weeks: number analyzed (Participants) | 56 | 64
  8 weeks | 30.11 (4.82) | 27.97 (5.15)
  3 month follow-up: number analyzed (Participants) | 51 | 59
  3 month follow-up | 30.73 (4.97) | 28.17 (6.14)
  6 month follow-up: number analyzed (Participants) | 47 | 52
  6 month follow-up | 31.13 (4.38) | 28.38 (5.72)

12. Secondary Outcome: The Behaviour Rating Inventory of Executive Function-Adult (BRIEF-A)
Description: The Behaviour Rating Inventory of Executive Function-Adult (BRIEF-A) is composed of 75 items within nine non-overlapping theoretically and empirically derived clinical scales. It has 2 broad indexes (Behavioural Regulation and Metacognition), an overall summary score, and three validity scales. This analysis examines the overall summary score. T scores (M = 50, SD = 10; transformations of the raw scale scores) are used to interpret the individual's level of executive functioning. Traditionally, T scores at or above 65 are considered clinically significant. Greater scores indicate greater deficits in executive functioning.
Time Frame: Change from Baseline to Week 8, 3 month follow up, 6 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t score
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
Number analyzed (Participants) | 63 | 69
t score
  Baseline: number analyzed (Participants) | 63 | 67
  Baseline | 60.37 (10.31) | 59.13 (11.28)
  8 weeks: number analyzed (Participants) | 59 | 64
  8 weeks | 51.14 (10.72) | 52.41 (11.30)
  3 month follow-up: number analyzed (Participants) | 54 | 61
  3 month follow-up | 50.13 (10.67) | 51.54 (11.08)
  6 month follow-up: number analyzed (Participants) | 52 | 57
  6 month follow-up | 50.65 (10.39) | 52.54 (13.60)

13. Secondary Outcome: The Work Productivity and Activity Impairment (WPAI)
Description: The WPAI questionnaire was developed for the purpose of collecting productivity loss data within clinical trials and is suitable for direct translation into a monetary figure. The WPAI yields four types of scores: 1. Absenteeism (work time missed) 2. Presenteesism (impairment at work / reduced on-the-job effectiveness) 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism) 4. Activity Impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: Change from Baseline to Week 8, 3 month follow up, 6 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of work productivity loss
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
Number analyzed (Participants) | 63 | 69
percentage of work productivity loss
  Baseline: number analyzed (Participants) | 26 | 22
  Baseline | 23.33 (34.04) | 18.28 (31.29)
  8 weeks: number analyzed (Participants) | 32 | 27
  8 weeks | 7.42 (21.48) | 11.54 (28.05)
  3 month follow-up: number analyzed (Participants) | 33 | 29
  3 month follow-up | 6.25 (20.14) | 5.85 (20.37)
  6 month follow-up: number analyzed (Participants) | 63 | 29
  6 month follow-up | 5.77 (19.36) | 5.63 (19.92)

14. Secondary Outcome: Credibility/Expectancy Questionnaire (CEQ)
Description: The Credibility/Expectancy Questionnaire (CEQ) is a 6-item questionnaire that captures both credibility beliefs and outcome expectancy. Questions on this scale are rated on a 1-to-9 point or 0-100% Likert scale, depending on the exact question. The scale was adapted to separately assess: (1) credibility beliefs for insomnia; (2) credibility beliefs for PCI; (3) expectancy beliefs for insomnia; and (4) expectancy beliefs for PCI. Since the CEQ utilizes two scales during the administration (1-9, and 0-100%), a composite score was derived for each factor (expectancy and credibility) by first standardizing the individual items and then summing those items for each factor yielding total scores, where higher values indicate stronger credibility and expectancy beliefs. Credibility beliefs scores ranged from 0 to 23 and expectancy beliefs scores ranged from 0 to 27.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
Number analyzed (Participants) | 63 | 69
scores on a scale
  Baseline credibility: number analyzed (Participants) | 63 | 68
  Baseline credibility | 15.37 (4.42) | 16.43 (3.94)
  Baseline expectancy: number analyzed (Participants) | 63 | 68
  Baseline expectancy | 19.68 (4.48) | 20.28 (4.19)

ADVERSE EVENTS:
Time Frame: 6 months
Description: We followed the CONSORT 2022 guidelines for reporting harms 33 to ensure that adverse events (AEs) were: (1) Clearly defined; (2) Clearly stated in measurement and methodology; (3) Reported with an attribution; (4) Reported with severity. Participants were asked about five categories of possible AEs: (1) Distress, illness, or incidents; (2) New development of symptoms; (3) Unplanned medical visits/procedures; (4) Unplanned need to take medication; (5) Any other physical/mental health concern.
Arm/Group | Cognitive Behaviour Therapy for Insomnia (CBT-I) | Waitlist Control Group
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/69
Serious Adverse Events (participants affected / at risk) | 2/63 | 2/69
Other Adverse Events (participants affected / at risk) | 12/63 | 14/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behaviour Therapy for Insomnia (CBT-I) (N=63) | Waitlist Control Group (N=69)
Infection (General disorders) | 1 (1) | 1 (1)
Surgery (General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behaviour Therapy for Insomnia (CBT-I) (N=63) | Waitlist Control Group (N=69)
Headache or Migraine (General disorders) | 4 (4) | 2 (2)
Increased Pain (General disorders) | 5 (5) | 7 (7) — (New occurrence of pain or flare up of existing pain; e.g., hip, joints, shoulder, back, neck, chest, muscle, etc.)
Fatigue (General disorders) | 3 (3) | 5 (5)

LIMITATIONS AND CAVEATS:
Clinical trials using a waitlist condition generally inflate treatment effects; Use of waitlist control precluded comparing groups on long-term outcomes; Close to half of the patients in this trial were long-term cancer survivors, which may reduce the ability to attribute their functioning to their cancer diagnosis or treatments; The improvements observed in cancer-related cognitive impairment are only generalizable to patients who have insomnia and cognitive impairment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/48/NCT04026048/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/48/NCT04026048/ICF_001.pdf